CLINICAL TRIAL: NCT00887809
Title: Phase II Trial Of Gemcitabine and Docetaxel With Bevacizumab in Selected Sarcoma Subtypes
Brief Title: Gemcitabine and Docetaxel With Bevacizumab in Selected Sarcoma Subtypes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-015
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Sarcoma; Leiomyosarcoma; Malignant Fibrous; Histiocytoma; Angiosarcoma
Keywords: Bevacizumab (avastin); Gemcitabine; Taxotere (docetaxel); 09-015; Soft tissue
MeSH Terms: conditions — Sarcoma; Leiomyosarcoma; Histiocytoma; Hemangiosarcoma | interventions — Gemcitabine; Docetaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gemcitabine and docetaxel with bevacizumab (Experimental): Patients will receive bevacizumab at 15 mg/kg on day 1 of each 21-day cycle intravenously over 30 minutes followed by a one hour (+30/-15 min) break. For cycles 1 through 6, gemcitabine will be administered at 900 mg/m2 over 90 minutes on day 1 and 8 of a 21-day cycle. Docetaxel will be administered at 75 mg/m2, over 60 minutes, on day 8. This will be followed by either 5 days of filgrastim or a single injection of pegfilgrastim. For cycles 7 and beyond, gemcitabine will be given at 800 mg/m2 over 30 minutes on day 1 and 8; docetaxel will be given at 35 mg/m2 over 30 minutes, also on days 1 and 8.
  Interventions: Drug: gemcitabine; Drug: docetaxel; Drug: bevacizumab

INTERVENTIONS:
Drug: gemcitabine
Drug: docetaxel
Drug: bevacizumab

SUMMARY:
The purpose of this study is to test whether an experimental drug called bevacizumab given together with gemcitabine and docetaxel, a standard chemotherapy regimen for sarcoma, can help sarcoma patients. This trial will examine what effects, good and/or bad the combination of gemcitabine, docetaxel and bevacizumab has on sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable metastatic or locally recurrent leiomyosarcoma, Malignant Fibrous Histiocytoma (MFH, also known as high grade Undifferentiated Pleomorphic Sarcoma) pleomorphic liposarcoma, rhabdomyosarcoma or angiosarcoma.
* Zero to one prior chemotherapy regimens for metastatic disease. Prior adjuvant therapy will not count provided it was more than one year previously.
* Measurable disease as defined by RECIST
* Adequate performance status - ECOG 0 or 1
* Patients must be recovered from the toxic effects of prior chemotherapy or radiation. Therapy may not start until at least 3 weeks since prior cytotoxic chemotherapy, two weeks from completion of radiation therapy, and one week for patients on tyrosine kinase inhibitors or other targeted therapy.
* Age 18 To 75. As it is quite difficult to administer high dose docetaxel with gemcitabine, to the elderly, in order to protect patient safety, we will restrict eligibility to patients between the ages of 18 and 75.
* Adequate hematologic, hepatic and renal function as defined below
* Hemoglobin > or = to 8.0 g/dl
* Absolute neutrophil count > or = to 1,500/mm3
* Platelet count > or = to 100,000/mm3
* Total Bilirubin < or = to1.5 x upper limit of normal (ULN).
* ALT (SGOT) or AST (SGPT) < or = to 5 x ULN.
* Alkaline Phosphatase < or = to 2.5 x ULN or ≤ 5 x ULN in presence of liver metastases.
* Serum creatinine 2.0 mg/dL
* Ability to understand informed consent and comply with treatment protocol
* Normal cardiac ejection fraction
* Urine protein:creatinine (UPC) ratio < than or = to 1.0 at screening

Exclusion Criteria:

* Uncontrolled intercurrent illness including infection or congestive heart failure within 6 months.
* Prior therapy with gemcitabine, docetaxel or bevacizumab
* Patients receiving other investigational agents
* Patients with known brain metastases
* Pregnancy or unwillingness to use effective birth control
* Patients with HIV disease will be permitted, only if they are on effective anti-retroviral therapy, have a CD4 count greater than 400, and have had no opportunistic infections within the past 6 months.
* Patients on anti-coagulation will be permitted if they are on a stable dose of warfarin or low-molecular weight heparin, and have had no major bleeds within the past 6 months.
* Inability to comply with study and/or follow-up procedures.
* Life expectancy of less than 12 weeks.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* Active malignancy, other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix within last three years
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg lasting > 24 hours on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection), requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, active ulcer, or non-healing bone fracture
* Proteinuria at screening as demonstrated by
* Urine protein:creatinine (UPC) ratio > or = to 1.0 at screening (patients discovered to have UPC ratio > or = to 1.0 at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of bevacizumab
* Pregnant (positive pregnancy test) or lactating. Use of effective means of contraception (men and women) in subjects of child-bearing potential
* History of hemoptysis (bright red blood of 1/2 teaspoon or more per episode) within 3 months prior to study enrollment.
* Any history of stroke or transient ischemic attack within 6 months
* History of myocardial infarction or unstable angina within 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-04; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Tap, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine, Docetaxel, Bevacizumab: Gemcitabine, Docetaxel, Bevacizumab
- Gemcitabine, Docetaxel, Placebo: Gemcitabine, Docetaxel, Placebo
Period: Overall Study
Arm/Group | Gemcitabine, Docetaxel, Bevacizumab | Gemcitabine, Docetaxel, Placebo
Started | 37 | 10
Completed | 33 | 10
Not Completed | 4 | 0
Not completed — Patient Not Treated | 3 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine, Docetaxel, Bevacizumab | Gemcitabine, Docetaxel, Placebo | Total
Number analyzed (Participants) | 37 | 10 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 7 | 33
  >=65 years | 11 | 3 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 2 | 24
  Male | 15 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: Overall Objective Response will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Gemcitabine, Docetaxel, Bevacizumab | Gemcitabine, Docetaxel, Placebo
Number analyzed (Participants) | 33 | 10
participants
  Complete Response (CR) | 0 | 1
  Partial Response (PR) | 9 | 1
  Stable Disease (SD) | 23 | 7
  Progression of Disease (POD) | 1 | 1

ADVERSE EVENTS:
Arm/Group | Gemcitabine, Docetaxel, Bevacizumab | Gemcitabine, Docetaxel, Placebo
Serious Adverse Events (participants affected / at risk) | 12/37 | 6/10
Other Adverse Events (participants affected / at risk) | 33/37 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Docetaxel, Bevacizumab (N=37) | Gemcitabine, Docetaxel, Placebo (N=10)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Death not assoc w CTCAE term- Death NOS (General disorders) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (General disorders) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hemorrhage/Bleeding, other (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Infection normal Absolute Neutrophil Counts/grade 1/2 neutrophils-Cellulitis(skin) (Infections and infestations) | 1 (1) | 0 (0)
Infection normal Absolute Neutrophil Counts/grade 1/2 neutrophils-Pneumonia(lung) (Infections and infestations) | 1 (1) | 0 (0)
Infection unknown Absolute Neutrophil Counts -Pneumonia(lung) (Infections and infestations) | 0 (0) | 1 (1)
Infection, other (Infections and infestations) | 2 (2) | 0 (0)
Leukocytes (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pain - Chest/thorax NOS (General disorders) | 1 (1) | 0 (0)
Pain - Extremity-limb (General disorders) | 1 (1) | 0 (0)
Pain - Pelvis (General disorders) | 0 (0) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Pulmonary/upper respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal/Genitourinary-Other (Renal and urinary disorders) | 0 (0) | 1 (1)
Syncope (fainting) (General disorders) | 1 (1) | 0 (0)
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Valvular heart disease (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Docetaxel, Bevacizumab (N=37) | Gemcitabine, Docetaxel, Placebo (N=10)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 19 (19) | 6 (6)
Alkaline phosphatase (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
ALT, SGPT (Blood and lymphatic system disorders) | 10 (10) | 3 (3)
AST, SGOT (Blood and lymphatic system disorders) | 10 (10) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Edema: limb (General disorders) | 3 (3) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (3) | 2 (2)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 17 (17) | 4 (4)
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 27 (27) | 8 (8)
Infection normal Absolute Neutrophil Counts/grade 1/2 neutrophils-Pneumonia(lung) (Infections and infestations) | 0 (0) | 1 (1)
International normalized ratio (INR) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 20 (20) | 5 (5)
Lymphopenia (Blood and lymphatic system disorders) | 16 (16) | 6 (6)
Magnesium, high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Mucositis (Clincal exam)- Oral cavity (General disorders) | 3 (3) | 0 (0)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 22 (22) | 5 (5)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 11 (11) | 3 (3)
Platelets (Blood and lymphatic system disorders) | 9 (9) | 3 (3)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Partial thromboplastin time (PTT) (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes